CLINICAL TRIAL: NCT03169803
Title: Cardiac Output Autonomic Stimulation Therapy for Acute Heart Failure (COAST-AHF) - System Design Study
Brief Title: Cardiac Output Autonomic Stimulation Therapy for Acute Heart Failure (COAST-AHF)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NeuroTronik Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 700022-01
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Heart Failure Acute
Keywords: Electrical Stimulation Therapy; Electrodes; Parasympathetic Nervous System; Sympathetic Fibers; Post Ganglionic; Congestive Heart Failure; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm, NeuroTronik CANS Therapy System (Experimental)
  Interventions: Device: NeuroTronik CANS Therapy™ System

INTERVENTIONS:
Device: NeuroTronik CANS Therapy™ System — The NeuroTronik CANS Therapy™ System is a percutaneous, catheter-based, bedside electrical stimulation system. The System consists of the single-use, disposable NeuroCatheter™ and NeuroCatheter™ Placement Kit, along with the reusable, bedside NeuroModulator™ Development System, and the NeuroTronik CANS Therapy™ Cable.

SUMMARY:
A feasibility study to investigate the safety and performance of the NeuroTronik Cardiac Autonomic Nerve Stimulation (CANS) Therapy System

DETAILED DESCRIPTION:
A single-arm, safety study intended to assess safety and system performance, and the feasibility to improve hemodynamics in patients with acute heart failure syndrome using transvenous, cardiac autonomic nerve stimulation (CANS) therapy. In addition, the effects of NeuroTronik CANS Therapy™ on the congestion of patients will be studied. The study proposes that the NeuroTronik CANS Therapy™ System be deployed during the acute heart failure syndrome hospital admission, along with existing standard treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Left Ventricular Ejection fraction < 40%, measured in the last year
2. At least two of the following:

   * Pulmonary Capillary Wedge Pressure > 18 mmHg
   * Pulmonary congestion on Chest X-ray
   * Jugular vein distension
   * Pulmonary rales
   * Edema
   * Dyspnea at rest
   * Two (2) emergency room visits or hospital admissions in the past three (3) months, or three (3) emergency room visits or admissions in the past six (6) months requiring intravenous diuretics, ultrafiltration or in-hospital inotropic therapy.
3. With or without evidence of low perfusion

Exclusion Criteria:

1. Systolic Blood Pressure < 90 mmHg or > 160 mmHg
2. Catecholamine or inotropic therapy within the previous 48 hours
3. Levosimendan within the previous 72 hours
4. Chronic outpatient catecholamine or inotropic therapy
5. Presence of implanted pacemaker, implantable cardioverter defibrillator or cardiac resynchronization therapy device
6. Presence of or prior vagal nerve stimulator
7. Coronary artery bypass graft surgery, percutaneous coronary intervention, acute myocardial infarction, or valve replacement within prior 1 month
8. Second or third degree heart block
9. History of atrial or ventricular arrhythmias
10. History of mitral or aortic valve stenosis or regurgitation
11. Hypertrophic obstructive or infiltrative cardiomyopathy
12. Prior vagotomy
13. Prior heart transplant
14. Narrow angle glaucoma
15. Renal failure - either on dialysis or serum creatinine > 2.0 mg/dl
16. Hepatic failure - bilirubin, serum glutamic oxaloacetic transaminase, or serum glutamic pyruvic transaminase > four times upper limit of normal
17. Life expectancy < 12 months per physician judgment
18. Women who are pregnant
19. Allergy to fentanyl, midazolam, propofol, eggs, egg products, soybeans, or soy products
20. Subjects unwilling or unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-05-19 (Actual); Primary Completion 2019-05-19 (Estimated); Study Completion 2019-06-19 (Estimated)

PRIMARY OUTCOMES:
Arterial blood pressure | 24 hours
Heart Rate | 24 hours

SECONDARY OUTCOMES:
Cardiac output | 24 hours
Pulmonary capillary wedge pressure | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Temístocles Díaz, MD, Principal Investigator — Hospital Punta Pacífica, Panama City, Panama
Locations (1):
- Hospital Punta Pacífica, Panama City, Panama

IPD SHARING:
Plan to Share IPD: Undecided